CLINICAL TRIAL: NCT01435707
Title: The Effect of Epidural Steroid Injections on Glycemic Control in Diabetic Patients According to the Doses of Steroids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Woo Seog Sim, Associate Professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2011-08-058
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Low Back Pain
Keywords: epidural steroid injection; triamcinolone; fasting blood glucose; diabetes mellitus
MeSH Terms: conditions — Low Back Pain; Diabetes Mellitus | interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Caudal 40 group (Experimental): subjects who undergo caudal epidural block with triamcinolone 40 mg
  Interventions: Other: epidural steroid injection with Triamcinolone 40mg
- STE 20 group (Experimental): subjects who undergo selective transforaminal block with triamcinolone 20 mg
  Interventions: Other: Selective transforaminal epidural block with triamcinolone 20 mg
- Caudal 20 mg (Experimental): subjects who undergo caudal epidural block with triamcinolone 20 mg
  Interventions: Other: caudal epidural steroid injection with Triamcinolone 20mg
- STE 40 group (Experimental): subjects who undergo selective transforaminal block with triamcinolone 40 mg
  Interventions: Other: Selective transforaminal epidural block with triamcinolone 40 mg

INTERVENTIONS:
Other: epidural steroid injection with Triamcinolone 40mg — epidural steroid injection with Triamcinolone 40mg
  Other Names: Triamcinolone; epidural steroid injection; caudal epidural block
  Arms: Caudal 40 group
Other: Selective transforaminal epidural block with triamcinolone 20 mg — Selective transforaminal epidural block with triamcinolone 20 mg
  Other Names: selective transforaminal block; Triamcinolone; epidural steroid injection
  Arms: STE 20 group
Other: caudal epidural steroid injection with Triamcinolone 20mg — caudal epidural steroid injection with Triamcinolone 20mg
  Other Names: Triamcinolone; epidural steroid injection; caudal epidural block
  Arms: Caudal 20 mg
Other: Selective transforaminal epidural block with triamcinolone 40 mg — Selective transforaminal epidural block with triamcinolone 40 mg
  Other Names: selective transforaminal block; Triamcinolone; epidural steroid injection
  Arms: STE 40 group

SUMMARY:
There has been no reports of the effect of various kinds of steroid or various dose of steroid which are commonly used in the clinical setting. Previous studies have simply shown that the blood glucose level is elevated in diabetes patients and did not show or suggest the adequate strategy of epidural steroid injection in diabetes patients regarding steroid type, dosage or injection interval. Therefore, the investigators tried to evaluate the effect of different dosage of triamcinolone, which is a commonly used steroid in epidural steroid injection, on the blood glucose level.

DETAILED DESCRIPTION:
It is well known that blood glucose level is elevated in diabetes patients more than non-diabetes patients who underwent the epidural steroid injection. However, there has been no reports of the effect of various kinds of steroid or various dose of steroid which are commonly used in the clinical setting. Previous studies have simply shown that the blood glucose level is elevated in diabetes patients and did not show or suggest the adequate strategy of epidural steroid injection in diabetes patients regarding steroid type, dosage or injection interval. Therefore, the investigators tried to evaluate the effect of different dosage of triamcinolone, which is a commonly used steroid in epidural steroid injection, on the blood glucose level.

ELIGIBILITY:
Inclusion Criteria:

* subjects who undergo epidural steroid injection (caudal epidural injection or selective transforaminal block) in the pain medicine outpatient clinic
* subjects older than 20 yrs.

Exclusion Criteria:

* ASA (American society of Anesthesiologists class) III or more
* severe cardiopulmonary disease or brain disorder
* Subjects diagnosed uncontrolled diabetes with complications
* subjects undergoing hormone therapy
* subjects with active infection
* subjects with pregnancy
* subjects with recent stress condition such as surgery or trauma
* subjects with active neurologic disorder
* those with anticoagulation therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
fasting blood glucose level | at 7:00 am of postprocedure day 1
  before breakfast (fasting state)
fasting blood glucose level | at 7:00 am of postprocedure day 2
  before breakfast (fasting state)
fasting blood glucose level | at 7:00 am of postprocedure day 3
fasting blood glucose level | at 7:00 am of postprocedure day 4
fasting blood glucose level | at 7:00 am of postprocedure day 5
fasting blood glucose level | at 7:00 am of postprocedure day 6
fasting blood glucose level | at 7:00 am of postprocedure day 7
fasting blood glucose | at 7:00 am of postprocedure day 14

SECONDARY OUTCOMES:
post-prandial glucose level | 2 hour after dinner at postprandial day 1, 2, 3, 4, 5, 6, 7, 14
  2 hour after dinner
visual analogue scale of subjective pain | at 7 p.m. of postprocedure day 1, 2, 3, 4, 5, 6, 7, 14
  at 7:00 am of postprocedure day 5

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim WH, Sim WS, Shin BS, Lee CJ, Jin HS, Lee JY, Roe HJ, Kim CS, Lee SM. Effects of two different doses of epidural steroid on blood glucose levels and pain control in patients with diabetes mellitus. Pain Physician. 2013 Nov-Dec;16(6):557-68. PMID 24284841